CLINICAL TRIAL: NCT06227065
Title: Precise Neoadjuvant Chemoresection of Low Grade NMIBC Guided by Drug Screens in Patient Derived Organoidst: A Single Center, Open-label, Phase II Trial
Brief Title: Precise Neoadjuvant Chemoresection of Low Grade NMIBC
Acronym: POLO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Spitalzentrum Biel (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZB-URO-24-001
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Bladder Cancer; Non-muscle Invasive Bladder Cancer; Low-risk
Keywords: Patient derived organoids; Neoadjuvant chemoresection; Precise drug selection
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Epirubicin; Mitomycin; Gemcitabine; Docetaxel

STUDY DESIGN:
Intervention Model Description: Phase II, all 28 patients will follow the same treatment. Only, selection of the use drug is performed using drug screens in patient derived organoids and is specific for each patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Epirubicin (Experimental): Patients in that PDOs show highest response to this drug in-vitro will be treated with Epirubicin.
  Interventions: Drug: Epirubicin
- Mitomycin (Experimental): Patients in that PDOs show highest response to this drug in-vitro will be treated with Mitomycin.
  Interventions: Drug: Mitomycin
- Gemcitabine (Experimental): Patients in that PDOs show highest response to this drug in-vitro will be treated with Gemcitabine.
  Interventions: Drug: Gemcitabine
- Docetaxel (Experimental): Patients in that PDOs show highest response to this drug in-vitro will be treated with Docetaxel.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Epirubicin — In PDOs from patients that show highest response to Epirubicin, this drug will be instilled intravesically once weekly for 6 times.
  Epirubicin will be used as a concentrate for injection/instillation 2 mg/ml in total 50mg per vial. Prior to use, the concentrate for injection is diluted with 25ml of 0.9% saline solution to obtain the final Solution with 1mg/ml of Epirubicin.
  Arms: Epirubicin
Drug: Mitomycin — In PDOs from patients that show highest response to Mitomycin, this drug will be instilled intravesically once weekly for 6 times.
  Mitomycin C will be used as 20mg dry powder. Prior to use, the powder will be dissolved in 50ml of 0.9% saline solution according to the manufacturer instructions
  Arms: Mitomycin
Drug: Gemcitabine — In PDOs from patients that show highest response to Gemcitabine, this drug will be instilled intravesically once weekly for 6 times.
  Gemcitabine will be used as 2000 mg/50ml. For intravesical application, 1000mg of gemcitabine (corresponding to 25ml) will be diluted in 25ml 0.9% saline solution, to obtain the gemcitabine concentration of 1000mg/50ml used for instillation.
  Arms: Gemcitabine
Drug: Docetaxel — In PDOs from patients that show highest response to Docetaxel, this drug will be instilled intravesically once weekly for 6 times.
  Docetaxel will be used as 140mg/7ml solution. For intravesical application, 48.825ml of saline will be added to 1.875ml Docetaxel solution (according 37.5mg of Docetaxel). The concentration of this solution is 0.74mg/ml by a total volume of the instillation solution of 50,7.
  Arms: Docetaxel

SUMMARY:
Based on the unmet clinical need to reduce invasiveness of treatment of low grade NMIBC, the investigators conduct this prospective, open label, single arm and single center phase II trial. The investigators aim to use drug screens in PDOs to guide neoadjuvant intravesical instillation therapy with either Epirubicin, Mitomycin C, Gemcitabine or Docetaxel to achieve chemoresection NMIBC.

DETAILED DESCRIPTION:
Bladder cancer is a disease of the elderly patient and related to several interventions and operations. Patients with a low risk non-muscle invasive bladder cancer (NMIBC) are treated by transurethral resection of the bladder tumor (TURBT). Due to the high recurrence rate of approximately 50% within 2 years of diagnosis, patients are followed in outpatient clinic by cystoscopy for at least 5 years.

Beside recurrence of low grade NMIBC to low grade disease, progression to higher grade or stage is infrequent to rare. Therefore, expectant management and actives surveillance seems to be an option for selected patients that are unfit for surgery. Moreover, intravesical chemoresection has been attempted in order to avoid surgery. However, all patients were treated with the same chemotherapeutic agent and anticipated response rates were missed.

At least four different drugs have been used in daily routine and/or clinical trials for instillation therapies in NMIBC. Namely, Epirubicin, Mitomycin C, Gemcitabine and Docetaxel have been investigated and administered.

The molecular landscape of NMIBC is heterogeneous. Not only the mutational pattern but also the transcriptomic characteristics vary between different NMIBC. Although different agents are used on a routine daily bases and in clinical trials, they have not been administered based on the molecular landscape or biological likelihood of response.

The investigators recently developed a pipeline for the generation of patient derived organoids (PDO) in NMIBC. In brief: The bladder cancer is sampled during TURBT. Generation of organoids has been carefully optimized in order to yield high viability from each sample. Beside confirmation of similarities of the molecular landscape between parental NMIBC and subsequent PDO (in approx. 30 samples), the investigators established a standardized protocol to perform drug screens on these PDOs.

In this trial (POLO Trial) the investigators aim to generate PDOs from bladder cancer biopsies that are harvested in the outpatient clinic. Subsequent drug screen in PDOs for Epirubicin, Mitomycin C, Gemcitabine and Docetaxel will identify the most effective agent in this given patient. Prior TURBT, patient will receive 6 intravesical instillations with the identified agent as neoadjuvant treatment in order to perform chemoresection of the tumor. Three months after initial diagnosis, TURBT will be performed as the standard treatment and to confirm response rate of precise chemoresection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed Informed Consent Form
* ECOG performance status of 0 or 1
* Previous history of low risk non-muscle invasive urothelial carcino-ma of the bladder with recurrent papillary tumor and negative urine cytology or Primary solitary papillary tumor, <3cm and negative urine cytology

Exclusion Criteria:

* Known previous high grade and/or intermediate or high risk non-muscle invasive bladder cancer
* Anticoagulation other than acetylsalicylic acid
* Previous Intravesical biological/immuno- (BCG) therapy
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Pathological response | 15 weeks
  Rate of patients that show complete pathological response to neoadjuvant chemoresection

SECONDARY OUTCOMES:
Number of patients with recurrence free survival | 1 Year
  Recurrence after neoadjuvant chemoresection and transurethral resection of the bladder tumor
Tolerability of instillation | 15 weeks
  Composite endpoint determined by standardized questionnaires (EORTC QLQ-C30, QLQ-NMIBC24 and IPSS)
Feasibility of drug screen | 4 weeks
  Rate of patients in which drug screen in patient derived organoids was successful

CONTACTS AND LOCATIONS:
Overall Officials: Roland Seiler, Prof., Study Chair — Spitalzentrum Biel, University of Bern
Locations (1):
- Roland Seiler, Biel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
After completion of the trial for the primary endpoint, deidentified data will be shared to other researches upon request.
Supporting Information: Study Protocol
Time Frame: After completion of the trial to the primary endpoint.